CLINICAL TRIAL: NCT02437825
Title: Prospective Randomized, Double-blind, Placebo-controlled Parallel Group Study of the Efficacy of Octreotide in Prevention of Salivary Fistulae After Post Radiation Salvage Surgery
Brief Title: Octreotide VS Placebo in Prevention of Salivary Fistulae After Post Radiation Salvage Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0102-15-HMO-CTIL
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2016-09

CONDITIONS: Fistula; Salivary Duct or Gland
MeSH Terms: conditions — Fistula | interventions — Octreotide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- octreotide treatment (Experimental): The studied drug Octreotide 100 mcg will be administered I.V in the evening prior to surgery and for two weeks on a thrice daily basis.
  Interventions: Drug: octreotide
- placebo treatment (Placebo Comparator): plasebo will be administrated I.V in the evening prior to surgery and two weeks on a thrice daily basis
  Interventions: Other: placebo

INTERVENTIONS:
Drug: octreotide — Octreotide has been in clinical use for thirty years and approved for use in Israel in acromegaly and functional gastroenteropancreatic tumours. It is currently being used extensively in surgical patients to prevent pancreatic fistulae1, and in lymphorrhea (both lymphatic malformations and leaks from the thoracic duct)
  Other Names: sundostatine
  Arms: octreotide treatment
Other: placebo — placebo ( saline) act as comperator in this study.
  Other Names: saline
  Arms: placebo treatment

SUMMARY:
Salivary fistulae have been the bane of surgical salvage in the era of primary chemoradiation for head and neck (H&N) cancers. The "blame"of prior chemoradiation tissue damage encouraged compensatory surgical techniques that focused on the insertion of non-irradiated tissue into the field. This study emphasizes a paradigm shift in the understanding and treatment of pharyngocutaneous fistulae. The detrimental effects of salivary enzymes on tissue healing and surgical anastomoses are addressed and novel treatment strategy is outlined.

DETAILED DESCRIPTION:
After signing an informed consent form, patients scheduled for total laryngectomy or for composite resections for oral/pharyngeal/laryngeal malignant tumors, will be randomly divided into two groups of about ten in each. The control group will receive a placebo while the study group will receive octreotide. All involved in the care of the patients and the patients themselves will be blinded to the drug given. The rest of the treatment will be equal in both groups and will adhere to the current departmental protocols in Otolaryngology/Oral-Maxillofacial Surgery.

The studied drug (Octreotide 100 mcg s/c) or placebo will be administered in the evening prior to surgery and subsequently for two weeks on a thrice daily basis.

Both groups will remain in hospital postoperatively for a minimum two week period (the current common practice). In addition to daily wound assessments, including daily grading of the pharyngocutaneous fistulae (using our grading system), the patients will also be evaluated for:

Serology:

1. Complete blood count and biochemistry including CRP and amylase will be assessed every 3 days.
2. GlucoChecks will be performed daily.

Imaging:

1. Patients will have an abdominal ultrasound to examine the gallbladder prior to and following completion of the two-weeks of therapy.

Admission stay:

Fistula prevention or acceleration of healing will be reflected in the admission time; generally, patients with fistulae suffer prolonged hospital stays.

Quality of Life Evaluation:

Evaluation of patients' quality of life will be based on two assessment scores:

1. Pain evaluation:

   Patients will rate their average head and neck region pain intensity with a 0-10 Numeric Rating Scale (NRS) (comprising 11 integers including 0), where 0 is "no pain" and 10 represent "the worst pain possible". Assessment will include a record of 'current NRS '-representing current pain and 'NRS maximum' representing maximal recalled pain in the in the last six months. The NRS highly correlates to other pain assessment scales and is a valid, reliable and easy to use tool in clinical dental practice.
2. Oral Health Impact Profile (OHIP-14) questionnaire:

The validated Hebrew version of the short OHIP (Oral Health Impact Profile) questionnaire (OHIP-14) will be used to assess the Oral health-related quality of life (OHRQoL). For each OHIP-14 question, subjects will be asked how frequently they had experienced the impact in the last six months. Responses will be made on a 5 point ordinal scale: 0-never , 1-hardly ever, 2-occasionally, 3- fairly often, and 4-very often. OHRQoL impairment will be characterized by the OHIP-14 global score, with a potential range of 0 (no adverse impacts within the last six months) to 56 (all 14 impacts experienced very often within the last six months). The OHIP-14 includes seven conceptual dimensions of oral health related quality of life. The dimensions are functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. OHIP-14 domains will be calculated for each of the domains by summing the response scores for the two corresponding items. Relationships between OHIP-14 score and various socio-demographic parameters, health-related behaviors and pain scores will be assessed among the study population.

CBCT sialography:

On order to monitor the progression of the salivary gland healing process a cone beam computorized tomography (CBCT) sialography will be implemented.

Saliva collection and analysis:

Patients from the 2 groups will be asked not to eat, drink or brush their teeth an hour before saliva collection. Thereafter, the saliva secretion rate from the affected parotid gland (in the operative side) will be measured between 8 to 12 AM using the Carlson-Crittenden collector. Prior to placement of the cup, the buccal mucosa will be dried with gauze and the Stensen's ducts will be slightly squeezed to locate the ducts' orifices. Salivary flow will be stimulated with 2% citric acid. Saliva will be collected for a total time of 5 minutes. Samples will be kept on ice during and after saliva collection. Thereafter, samples will be centrifuged at 14,000 rpm for 20 min at 4°C. Supernatant will collected and protein concentration will be determined according to Bradford (Bio-Rad, Hercules, CA, USA). Several components secreted in saliva will be assessed including: Cortisolamylase, cytokines, growth factors, elastases and proteinases. Octreotide levels in saliva will also be assessed. In addition, sialochemical analysis of Na+, K+, Cl-, Ca2+, PO43-, Mg2+ concentrations will be performed.

Proteomic analysis:

Depending on protein concentrations further analysis may include supplementary characterization of salivary biomarkers including SDS-PAGE analysis, two-dimensional analytical gels, mass spectrometry identification and database searching.

Statistics Numerical variables will be presented as means and standard deviations, while categorized variables will be presented as frequencies and percentages. A Pearson's correlation coefficient method will be used. Differences between variables will be subjected to univariate analysis by t-test and ANOVA. The statistical processing will be established by SPSS 21.0. Statistical level of significance chosen as P < 0.05.

To examine the factors associated OHIP-14 total score in a multivariate model a conceptual hierarchical multiple regression model will be adopted within the uni-variate data7. This well-established approach employs sequential adjustments from distal to proximal determinants of a health condition, with the aim of elucidating their relationships. Conceptual analysis, contrary to statistical decisions on significant determinants of diseases, adopts a theoretical ordering. The ordering of variables is conceptually determined in accordance with the hypothesis which assumes which variables have confounding effects, and which variables have a modification effect.

ELIGIBILITY:
Inclusion Criteria:

* Chemoradiation
* Total laryngectomy
* Composite resections for oral/pharyngeal/laryngeal malignant tumors

Exclusion Criteria:

* Pregnancy
* Patients with malabsorption syndrome, short bowel or chologenic diarrhea not controlled by specific therapeutic means
* Patients with uncontrolled diabetes mellitus or a fasting plasma glucose > 250mg/d

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
elimination of post-radiation salivary fistulae | up to 7 days after the surgery
  yes/no fistulae formation

SECONDARY OUTCOMES:
saliva secretion rate | up 14 days after the surgery
  saliva collection
pain evaluation | up to 14 days after the surgery
  using of Numeric Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: jeffrey weinberger, MD, Principal Investigator — hadassah MO
Locations (1):
- HadassahMO, Jerusalem, Israel

REFERENCES:
- [Background] Gilbert MR, Sturm JJ, Gooding WE, Johnson JT, Kim S. Pectoralis major myofascial onlay and myocutaneous flaps and pharyngocutaneous fistula in salvage laryngectomy. Laryngoscope. 2014 Dec;124(12):2680-6. doi: 10.1002/lary.24796. Epub 2014 Jul 30. PMID 25132580
- [Background] Agra IM, Carvalho AL, Pontes E, Campos OD, Ulbrich FS, Magrin J, Kowalski LP. Postoperative complications after en bloc salvage surgery for head and neck cancer. Arch Otolaryngol Head Neck Surg. 2003 Dec;129(12):1317-21. doi: 10.1001/archotol.129.12.1317. PMID 14676158
- [Background] Bomeli SR, Desai SC, Johnson JT, Walvekar RR. Management of salivary flow in head and neck cancer patients--a systematic review. Oral Oncol. 2008 Nov;44(11):1000-8. doi: 10.1016/j.oraloncology.2008.02.007. Epub 2008 May 16. PMID 18486528
- [Background] Loguercio C, de Sio I, Romano M, del Vecchio Blanco C, Coltorti M. Effect of somatostatin on salivary secretion in man. Digestion. 1987;36(2):91-5. doi: 10.1159/000199405. PMID 2436964
- [Background] Spinell C, Ricci E, Berti P, Miccoli P. Postoperative salivary fistula: therapeutic action of octreotide. Surgery. 1995 Jan;117(1):117-8. doi: 10.1016/s0039-6060(05)80242-9. No abstract available. PMID 7809829
- [Background] Victora CG, Huttly SR, Fuchs SC, Olinto MT. The role of conceptual frameworks in epidemiological analysis: a hierarchical approach. Int J Epidemiol. 1997 Feb;26(1):224-7. doi: 10.1093/ije/26.1.224. PMID 9126524